CLINICAL TRIAL: NCT06204185
Title: Clinical and Biochemical Evaluation of the Use of Locally Delivered Metformin as an Adjunctive Therapy to Non Surgical Periodontal Treatment of Periodontitis Patients (Randomized Controlled Study)
Brief Title: Clinical and Biochemical Evaluation of 1% Metformin in Non-surgical Treatment of Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sameh Mohamed Magdy Abou El-Kheir, Assistant Lecturer - Faculty of Dentistry - Delta University for Science and Technology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FD-ASUREC.IM011967
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Evaluate the clinical parameters ( Probing Depth, Clinical Attachment Level, Gingival and Plaque Indices) before & after the application of locally delivered metformin as an adjunctive therapy to non surgical periodontal treatment of Stage III periodontitis.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1% Metformin (Active Comparator): 1% Metformin Delivered in biodegradable gel. Frequency- One dose each at baseline, 3 months and 6 months.
  Interventions: Drug: Metformin
- Control Group (Placebo Comparator): Placebo gel without the active ingredient. Delivered in biodegradable gel. Frequency- One dose each at baseline, 3 months and 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Locally delivered Metformin gel in the treatment of periodontitis patients
  Arms: 1% Metformin
Drug: Placebo — Placebo gel consist of drug without the active component.
  Arms: Control Group

SUMMARY:
The aim of the study to evaluate the clinical and biochemical efficacy of 1% Metformin gel in treatment of periodontitis patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage III Grade A Periodontitis.
* Systemically free according to the modified Burkitt's health history questionnaire, Group I. (Glick et al., 2021).
* Good compliance with the plaque control instructions following initial therapy.
* Availability for follow up and maintenance program.

Exclusion Criteria:

* Smokers
* Pregnant and lactating females.
* Vulnerable groups of patients' e.g (prisoners, handicapped patients and decisionally impaired individuals).

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
RANKL and Osteoprotegrin levels in Gingival Crevicular Fluid before & after application of metformin as an adjunctive therapy to non surgical periodontal treatment of Stage III periodontitis. | Baseline and 1 month after the gel application

SECONDARY OUTCOMES:
Plaque index (PI) | Baseline, 3 Months and 6 Months post operatively.
Gingival Index (GI) | Baseline, 3 Months and 6 Months post operatively.
Probing depth (PD) | Baseline, 3 Months and 6 Months post operatively.
Clinical attachment level (CAL) | Baseline, 3 Months and 6 Months post operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Sameh Magdy Abou El-Kheir, Cairo, Egypt

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT06204185/Prot_SAP_000.pdf